CLINICAL TRIAL: NCT03742427
Title: Effect of Cervical Collar on the Optic Nerve Sheath in Minor Head Trauma Patients
Brief Title: Effect of Cervical Collar on the Optic Nerve Sheath Diameter in Minor Head Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09.2018.298
Record Dates: First submitted 2018-09-25; First posted 2018-11-15 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Head Trauma
Keywords: ultrasonography; optic nerve sheath; head trauma
MeSH Terms: conditions — Craniocerebral Trauma | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- effect of c-collar in optic nerve sheath diameter (Experimental): Comparing the effect of c-collar in minor head trauma patients by using optic nerve sheath diameter ultrasonography
  Interventions: Diagnostic Test: ultrasonography

INTERVENTIONS:
Diagnostic Test: ultrasonography — optic nerve sheath diameter measurement will be done by ultrasonography on both eyes

SUMMARY:
This is randomized, controlled and blinded study was performed in minor head trauma patients. Two sonographers measured optic nerve sheath diameters (ONSD) of each subjects' eyes separately for different time points. Then a mean ONSD was calculated for before c-collar placement (T0), 5 and 20 minutes in supine position.

DETAILED DESCRIPTION:
Head trauma is an important cause of morbidity and mortality. Increased intracranial pressure (ICP) can lead to decreased cerebral perfusion and tissue damage. It is important to be able to detect increased ICP on time, so that treatment can be initiated to prevent further brain damage. The measurement of optic nerve sheath diameter (ONSD) has been proposed as a non-invasive and rapid way to assess elevated ICP (1-2). Traditional ICP monitoring methods such as external ventricular devices are invasive and time-consuming and can only be performed by trained personnel at trauma centers.

The optic nerve is surrounded by a protective sheath and is found on the back of the globe. Easily evaluated with ultrasonics. This is typically done with a linear probe measuring the diameter of the optic nerve sheath 3 mm back from where the contrast is highest. The normal upper limit for adults is 5 mm, the values above are considered abnormal. Many studies have shown that an increased ONSD measured by bedside ultrasound correlates with increased IDC and in one study there is a correlation between ONSD> 5 mm and ICP> 20 cm H2O.

Cervical spine (c-arms) and cervical vertebrae are often temporarily immobilized in patients with head trauma. It has been shown that placement of c-arms increases IBP. The decrease in venous outflow caused by c-arms in the forehead is an important mechanism for this increase in ICP. The increase in ICP occurs simultaneously with the application of c-arms in cadaver. It is thought that increased ONSD in trauma patients may be related to c-arms.

If a c-collar application is found to increase ONSD, this trauma may make it difficult to use ONSD as an non-invasive estimate of ICP in patients.

To the best of our knowledge, there is a study in healthy individuals investigating the possible effect of c-collar administration on ONSD. However, there is no comparative study of patients with head trauma. The investigators tried to measure ONSD before and after placement of cervical limbs in cases with minor head trauma. The aim of our study is to identify changes in the optic nerve sheath measurement after placement of the c-arms, and to determine whether these changes are due to the time immobilized by the c-arms.

This is randomized, controlled and blinded study was performed in minor head trauma patients. Two sonographers measured optic nerve sheath diameters (ONSD) of each subjects' eyes separately for different time points. Then a mean ONSD was calculated for before c-collar placement (T0), 5 and 20 minutes in supine position.

ELIGIBILITY:
Inclusion Criteria:

* Patients with minor head trauma
* Patients over 18 years and under 65 years
* Those who signed the Informed Consent Form

Exclusion Criteria:

* Patients who can not be followed for any reason (treatment, refusal, unauthorized leave, referral to the center, etc.)
* Patients who withdraw their consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-05-06 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sinan Karacabey, Study Director — Marmara University
Locations (1):
- Sinan Karacabey, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Woster CM, Zwank MD, Pasquarella JR, Wewerka SS, Anderson JP, Greupner JT, Motalib S. Placement of a cervical collar increases the optic nerve sheath diameter in healthy adults. Am J Emerg Med. 2018 Mar;36(3):430-434. doi: 10.1016/j.ajem.2017.08.051. Epub 2017 Aug 26. PMID 28865838
- [Background] Maissan IM, Ketelaars R, Vlottes B, Hoeks SE, den Hartog D, Stolker RJ. Increase in intracranial pressure by application of a rigid cervical collar: a pilot study in healthy volunteers. Eur J Emerg Med. 2018 Dec;25(6):e24-e28. doi: 10.1097/MEJ.0000000000000490. PMID 28727580

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Effect of C-collar in Optic Nerve Sheath Diameter
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Effect of C-collar in Optic Nerve Sheath Diameter
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.44 (6.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 50
Optic Nerve Sheath Diameter [Mean (Standard Deviation); unit: milimeters] — These measurements are the baseline measurements of the patients at time point "0" when they appeal to the emergency department before c-collar application.
  milimeters | 4.71 (0.22)

OUTCOME MEASURES:

1. Primary Outcome: Sonographic Evaluation of Cervical Collar Effects on the Optic Nerve Sheath Diameter in Head Trauma Patients
Description: We hypothesised that optic nerve sheath diameter raises after c-collar application in minor head trauma patients
Time Frame: 20 minutes
Measure: Mean (Standard Deviation); unit: Milimeter
Arm/Group | Effect of C-collar in Optic Nerve Sheath Diameter
Number analyzed (Participants) | 50
Milimeter
  0th Minute | 4.71 (0.22)
  5th minute | 5.19 (0.41)
  20th minute | 5.26 (0.45)

ADVERSE EVENTS:
Time Frame: 1 hour from appealing to emergency department
Description: No serious adverse events (death) or other adverse events (pain, hypotension, loss of vision ) were observed till the time frame due to study.
Arm/Group | Effect of C-collar in Optic Nerve Sheath Diameter
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/27/NCT03742427/Prot_SAP_000.pdf